CLINICAL TRIAL: NCT05660317
Title: Tip Control Assessment to Determine the Accuracy of Snare Tip Soft Coagulation to the Margin of Defects After EMR Predicts Polypectomy Experience and Procedural Difficulty
Brief Title: Assessment of Endoscopic Tip Control Using a Novel Score Based on the Snare Tip Soft Coagulation of Polypectomy Margin Defects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2022-0178
Record Dates: First submitted 2022-12-02; First posted 2022-12-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Polyp
Keywords: Endoscopy; Training; Polypectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Tip control score — Scoring of endoscopist's tip control performing snare tip soft coagulation to the margins of a endoscopic mucosal resection (EMR) defect

SUMMARY:
Colorectal cancer is the third most common malignancy worldwide and the second leading cause of cancer related death with approximately 880 792 deaths every year (9,2% of the global yearly 9.6 million cancer deaths). Screening for polyps is done by colonoscopy, which is considered the gold standard for screening and removal of polyps and has been proven to reduce the global colorectal cancer burden significantly. Endoscopic removal of polyps is preferred because of its efficiency, cost-effectiveness, and safety in comparison to surgery.

Endoscopic tip control is a fundamental component of high quality endoscopy. Endoscopic procedures are complex processes where cognitive processing and motoric output need to be perfectly aligned. This is reflected in endoscopic tip control. It is indispensable in every step of endoscopy: during insertion of the endoscope, where the tip of the endoscope needs to reach the caecum/terminal ileum/duodenum, without discomfort for the patient if under light sedation, during withdrawal of the endoscope in order not to miss any lesions, and also during every endoscopic treatment whether it is a simple polypectomy or a complex therapeutic procedure performed by expert endoscopists.

However, there is currently no tool available to assess endoscopic tip control. And very little is known about educating it.

The investigators developed a new, web-based scoring system to assess tip control. The intent of this study is to validate this novel tool so it can be used to assess endoscopists and evaluate their progress when training in endoscopy.

This study takes place at the University Hospital Ghent, which is a tertiary care center for gastrointestinal endoscopy. The investigators will validate the tool in this study, through assessment of endoscopists of varying experience while they use a technique of snare tip soft coagulation on the margin of a polypectomy defect. This technique has proven its use in preventing recurrence after polypectomy. The technique uses the tip of a snare (used to resect polyps) to deliver thermal energy to the margin of a polypectomy, also called margin ablation. Thermal energy is applied by a hit on a pedal (operated with the foot), every hit needs to be exactly on the margin of the defect (not in the defect, not on normal mucosa around the defect). This requires a very steady and controlled handling of the endoscope and is an ideal technique to assess endoscopist's tip control. The score system will calculate the accuracy (number of correct hits over number of wrong hits) of tip control per second.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopists who perform endoscopic mucosal resections (EMR) at the University Hospital of Ghent, Belgium (UZ Gent)
* Patients, > 18 years of age, referred for EMR needing snare tip soft coagulation of the defect margins.

Exclusion Criteria:

* Endoscopists who do not consent to the study
* Patients who do not consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Endoscopists: all endoscopist (varying experience) performing polypectomy at the University Hospital of Ghent, Belgium (UZ Gent)
  Patients: all patients undergoing endoscopic mucosal resection of colorectal polyps
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Endoscopists' accuracy of tip control using a novel scoring system. | Through study completion, an average of 1 year (no intervention, the participant gets scored with every margin ablation he does)
  Assessment of the tip control accuracy of endoscopists with varying experience using a novel scoring system.
  The scoring system reports accuracy of tip control: correct hits/total hits (range of accuracy 0-100% with 0% no correct hits, and 100% best possible accuracy) and correct hits per second, where a high score demonstrates good accuracy in short period of time (participants is good en fast).

SECONDARY OUTCOMES:
Assessment of quality parameters of the novel tip control scoring system. | Through study completion, an average of 1 year
  Assess if the scoring system is user friendly and assess if it is feasable to use it in an endoscopy setting.
  * questions: was this score easy to use?
  * did you find it useful?
  * you feel we can improve? how? (free text box)

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Gent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No